# INFORMATIE- EN TOESTEMMINGSFORMULIER TOT DEELNAME AAN DE STUDIE

Versie 2 – 24 januari 2025

## Het Rufaida project: Onderzoek naar de impact van Ramadan vasten op het darm en vaginale microbioom

Onderzoekstudie aan de Universiteit Antwerpen, Faculteit Wetenschappen, Departement Bioingenieurswetenschappen en de Faculteit Geneeskunde en Gezondheidswetenschappen

#### I. Noodzakelijke informatie voor uw beslissing om deel te nemen

Beste deelnemer,

U wordt uitgenodigd om deel te nemen aan een onderzoek dat zich richt op het begrijpen van de interactie tussen de darm- en vaginale microbiomen door de effecten van het vasten tijdens de Ramadan te onderzoeken. Dit onderzoek is onderdeel van een bredere studie naar de impact van dieet en levensstijl op de vrouwelijke gezondheid, met speciale aandacht voor de microorganismen die in en op ons lichaam leven.

De afgelopen jaren is er steeds meer aandacht voor het menselijk microbioom (verzameling van micro-organismen, meer bepaald bacteriën, schimmels, gisten en virussen) en de rol die het speelt in onze gezondheid. Hoewel veel van deze studies zich hebben gericht op de microorganismen in de darm, is de interactie tussen de darm- en vaginale microbiomen nog onvoldoende onderzocht. Dit is bijzonder relevant voor vrouwen, aangezien een gezond vaginaal milieu cruciaal is voor hun algemene welzijn.

In onze eerdere studies, waaronder het Isala-project, hebben we aangetoond dat er significante linken bestaan tussen de samenstelling van de verschillende micro-organismen in van de darmen en de vagina. Dit onderzoek wil deze hypothese verder verkennen door te kijken naar de effecten van Ramadan vasten op deze microbiomen. We willen onderzoeken of het vasten, dat meestal gepaard gaat met een verandering in dieet en eetpatronen, invloed kan hebben op de hoeveelheid micro-organismen en het aantal verschillende soorten van deze microorganismen op één plek in zowel de darm als de vagina.

Voordat u beslist om deel te nemen, willen we u graag voorzien van gedetailleerde informatie over de studie, de mogelijke voordelen en risico's, en wat deelname voor u inhoudt. Dit proces staat bekend als "geïnformeerde toestemming."

Wij vragen u om de volgende pagina's aandachtig door te nemen. Mocht u vragen hebben, aarzel dan niet om contact op te nemen met de verantwoordelijke onderzoekers. Dit document is opgedeeld in drie delen: essentiële informatie om een weloverwogen beslissing te nemen, een sectie voor uw schriftelijke toestemming en bijlagen met aanvullende details over de studie.

Wij danken u voor uw interesse in ons onderzoek en hopen dat u ons zult helpen om meer te leren over de complexe relatie tussen dieet, microbiomen en de gezondheid van vrouwen.

#### 1. Als u aan deze klinische studie deelneemt, dient u het volgende te weten:

- Deze klinische studie wordt opgestart na evaluatie door het Ethisch Comité UZA/UA.
- De deelname is vrijwillig. Voor deelname is uw ondertekende toestemming nodig. Ook nadat u hebt getekend, kan u op elk moment de arts-onderzoeker laten weten dat u de deelname wilt stopzetten. De beslissing om al dan niet (verder) deel te nemen zal geen enkele negatieve invloed hebben op de kwaliteit van de zorgen noch op de relatie met de behandelende arts(en).
- De gegevens die in het kader van uw de deelname worden verzameld, zijn vertrouwelijk. Bij de publicatie van de resultaten is uw anonimiteit verzekerd.
- Er worden u geen kosten aangerekend voor specifieke behandelingen, bezoeken/consultaties, onderzoeken in het kader van deze studie.
- Indien u extra informatie wenst, kan u altijd contact opnemen met de verantwoordelijken van de studie (ondertekenden van dit document).

Aanvullende informatie over "Rechten van de deelnemer aan een klinische studie" vindt u in bijlage.

#### 2. Doelstelling en beschrijving van het studieprotocol

Met deze studie willen we u vragen om toestemming te geven voor deelname aan ons onderzoek naar de effecten van Ramadan-vasten op de samenstelling van micro-organismen in de darmen en vagina van gezonde Moslimvrouwen die zich niet in de menopauze bevinden, 18 jaar of ouder zijn, en die in Vlaanderen of Brussel wonen. Dit onderzoek beoogt een duur van acht weken, waarin we de impact van Ramadan-vasten op de microbiomen van zowel de darm als de vagina zullen bestuderen. In deze studie kan u ervoor kiezen om stalen af te nemen en de vragenlijsten in te vullen (studiegroep 1), of enkel de vragenlijsten in te vullen (studiegroep 2).

Deelnemers van studiegroep 1 zullen gedurende deze periode stoelgang en vaginale stalen zelf verzamelen, wekelijks éénmalig voorafgaand aan, tijdens, en na de Ramadan. Het onderzoek is opgezet als een studie over een langere periode, waarbij start gegevens zonder vasten worden verzameld gedurende de eerste twee weken, gevolgd door vier weken van vasten, en een eind periode van twee weken waar het normale eetritme wordt hersteld. Dit ontwerp stelt ons in staat om veranderingen binnen een individu te analyseren en de effecten van de dieetverandering die tijdens de Ramadan plaatsvindt, in kaart te brengen.

Het belang van dit onderzoek bestaat uit twee delen. Ten eerste willen we de onderzoeksvraag bestuderen dat Ramadan-vasten de omzetting van bepaalde suikers tot kleinere stoffen uit bepaalde darmbacteriën stimuleert, wat mogelijk leidt tot een verhoogde aanwezigheid van gunstige bacteriën in de vagina. Ten tweede willen we inzicht verkrijgen in hoe dieetpatronen, zoals vasten, de interactie tussen de darm- en vaginale microbiomen beïnvloeden, wat wijst op een link tussen de vagina en darm (ook wel de vagina-darm as genoemd).

Eerdere studies hebben aangetoond dat vasten de diversiteit en samenstelling van de verschillende darmbacteriën kan beïnvloeden, maar onderzoek naar de effecten van dieet op de vaginale micro-organismen blijft beperkt. Onze studie zal bijdragen aan het begrijpen van deze interacties en kan belangrijke implicaties hebben voor de gezondheid van vrouwen, vooral voor degenen die geïnteresseerd zijn in levensstijl- en dieetadviezen gebaseerd op

wetenschappelijke onderzoeken in plaats van medicamenteuze behandelingen voor vaginale klachten.

Indien u verkiest om enkele vragenlijsten in te vullen en geen vaginale en stoelgang stalen te nemen, dan kan u deelnemen in studiegroep 2. De deelnemers van zowel studiegroep 1 als groep 2 zullen gedurende de studie gevraagd worden om wekelijks een korte vragenlijst in te vullen om hun dieet en gezondheid te monitoren, waardoor we een gedetailleerd overzicht krijgen van de mogelijke veranderingen in samenstelling van micro-organismen en het totaal van alle chemische stoffen die ons lichaam produceert tijdens de stofwisseling. De verzamelde gegevens zullen worden geanalyseerd met behulp van geavanceerde statistische en bioinformatica-methoden. Wij hopen dat deze studie niet alleen bijdraagt aan de wetenschappelijke literatuur over micro-organismen op en in het menselijk lichaam, maar ook direct inzicht biedt aan de deelnemers over de samenstelling van deze micro-organismen van hun eigen lichaam en de invloed van hun dieet op hun gezondheid.

## 3. Verloop van de studie

De microbioomonderzoeken worden uitgevoerd aan de UAntwerpen, binnen het departement Bio-ingenieurswetenschappen in het Laboratorium van Toegepaste Microbiologie en Biotechnologie onder leiding van Prof. Dr. Ir. Sarah Lebeer. Het verloop van de studie is schematisch weergegeven in Figuur 1.



Figuur 1: Verloop van de studie.

Voorafgaand aan de studie zal een preselectiestap plaatsvinden. U wordt gevraagd om enkele vragen te beantwoorden die nagaat of u voldoet aan de inclusie- en exclusiecriteria, waaronder een evaluatie van uw gezondheidstoestand. Indien u wordt geselecteerd, zal uw deelname aan de studie acht weken in beslag nemen. Er wordt u gevraagd of u stalen wenst af te nemen of niet. Afhankelijk van uw antwoord wordt u in studiegroep 1 (wel stalen afnemen), of studiegroep 2 (geen stalen afnemen) geplaatst. De eerste vragenlijst zal ongeveer 35 minuten duren om in te vullen. De andere vragenlijsten zullen ongeveer 25 minuten in beslag nemen.

Voor studiegroep één die vaginale en stoelgang stalen zullen afnemen.

De eerste staalname vindt plaats één week voor de aanvang van de Ramadan (tijdspunt 1), waar u ook informatie ontvangt over het gebruik van de benodigde stalen en vragenlijsten. Na het afnemen van deze stalen komt u deze inleveren. Het tweede tijdspunt is enkele dagen voor de Ramadan (tijdspunt 2), gevolgd door een derde staalafname op tijdspunt 3. Na het afnemen van deze stalen komt u deze van tijdspunt 2 en 3 inleveren. Het vierde en vijfde tijdspunt zijn gedurende de Ramadan. Na het afnemen van de stalen komt u deze van tijdspunt 4 en 5 inleveren. De zesde staalname neemt u af op het einde van de Ramadan, gevolgd door de zevende staalafname vlak na het einde van de Ramadan en de achtste staalafname een week na de Ramadan. Na het afnemen van de stalen komt u deze van tijdspunt 6, 7 en 8 inleveren. Ieder tijdspunt wordt gepaard met een uitgebreide vragenlijst over algemene gezondheid, leefomgeving, mentale gezondheid, vaginale gezondheid, seksuele gezondheid en darm gezondheid.

Bij elk tijdspunt wordt u gevraagd om (thuis) één vaginale staal en één stoelgang staal af te nemen, met het doeleind voor het isoleren van hetDNA van de micro-organismen. Na het afnemen van de stalen moeten deze direct bewaard worden in de diepvriezer (ongeveer -20°C). Daarna moeten deze afgegeven worden in het lab van Prof. Sarah Lebeer (Campus Groenenborger, gebouw V, verdieping 5, adres: Groenenborgerlaan 171, 2020 Antwerpen).

Bij tijdspunt 1, 3, 5 en 8 wordt u gevraagd om (thuis) één additionele vaginale en één additionele stoelgang staal af te nemen, deze worden gebruikt om te achterhalen welke extra stoffen de aanwezige micro-organismen maken. Na het afnemen van de stalen moeten deze direct bewaard worden in de diepvriezer (ongeveer -20°C). Daarna moeten deze afgegeven worden in het lab van Prof. Sarah Lebeer (Campus Groenenborger, gebouw V, verdieping 5, adres: Groenenborgerlaan 171, 2020 Antwerpen).

Voor studiegroep twee (n=300) die enkel vragenlijsten zullen invullen.

Op elk tijdspunt zal u een mail krijgen met een vragenlijst over algemene gezondheid, leefomgeving, mentale gezondheid, vaginale gezondheid, seksuele gezondheid en darm gezondheid

De verwerking en analyse van de stalen zal plaatsvinden onder leiding van de UAntwerpen, binnen het departement Bio-ingenieurswetenschappen in het labo van Prof. Sarah Lebeer. We zullen het genetisch materiaal van de micro-organismen uit de stoelgang en vaginale stalen isoleren en kijken naar welke stoffen geproduceerd door de micro-organismen aanwezig zijn. Dit helpt ons om de algemene gezondheid te begrijpen en hoe de darm- en vaginale microbiomen met elkaar samenwerken.

Door deze gestructureerde aanpak hopen we inzicht te krijgen in de impact van Ramadan vasten op de micro-organismenmicro-organismen die aanwezig zijn in de darmen en de vagina, en welke gevolgen dit kan hebben voor de gezondheid van vrouwen. Na het aflopen van de studie zal je van ons een analyse krijgen van jouw persoonlijk microbioom met een woordje uitleg over de micro-organismen die we hebben gevonden. Op een later tijdstip zal er ook een algemene communicatie zijn over de resultaten van de studie. Indien je deze informatie niet wilt ontvangen kan je contact met ons opnemen.

**Met opmerkingen [SA1]:** Alles veranderen naar stoelgangstalen? Is misschien nog gemakkelijker

#### 4. Mogelijke risico's en ongemakken

Er is weinig tot geen risico of ongemak verbonden aan het verzamelen van de vaginale of stoelgang stalen.

De studie is goedgekeurd door de onafhankelijke Ethische Commissie van het Universitair Ziekenhuis Antwerpen en de Universiteit Antwerpen. Alle vrijwilligers zijn verzekerd volgens artikel 29 van de wet van 7 mei 2004 (UZA verzekeringscontract). De haalbaarheid, het belang, de veiligheid en de overeenstemming met de internationale aanbevelingen werden door deze Commissie geëvalueerd.

#### Voordelen van de studie

De onderzoeken zijn gemakkelijk uit te voeren en doen geen pijn. U helpt het onderzoek naar een verbeterde kennis omtrent de vrouwelijke gezondheid, alsook de gezondheid van hun eventuele partners en kinderen. Dit onderzoek bevordert ook de ontwikkeling van nieuwe gezondheidsbevorderende producten, onder andere ook producten op de basis van goede micro-organismen die bijdragen aan onze gezondheid.

#### Kosten en vergoeding

Voor de deelname aan deze studie zullen geen kosten gerekend worden voor de vrijwilligers aangezien alle diensten gratis zijn. Er zal geen financiële vergoeding voor de vrijwilligers voorzien worden. Er zal echter wel een Isala goodiebag met verschillende communicatie hulpmiddelen voorzien worden voor alle vrijwilligers om meer te leren over de vrouwelijke en intieme gezondheid en om het taboe hierrond te verbreken.

## 5. Vrijwillige deelname/ Intrekking van deelname uit de studie

U neemt vrijwillig deel aan de studie. U kan ook beslissen om niet aan het onderzoek deel te nemen en u kan op ieder moment uit het onderzoek stappen, zelfs als u dit formulier getekend heeft. Dit kan u doen door schriftelijk (via e-mail of brief) contact op te nemen met de hoofdonderzoekers. U kan vragen dat alle stalen die u gegeven heeft, vernietigd worden. De resultaten die op basis van uw stalen werden verkregen voordat u uw toestemming tot deelname hebt ingetrokken, blijven eigendom van de opdrachtgever.

#### 6. Biologische stalen die tijdens de studie worden afgenomen

De opdrachtgever van de studie verbindt zich ertoe dat de stalen uitsluitend gebruikt zullen worden in de context vermeld in de rubriek "verloop van de studie".

#### Stalen die voor de studieanalyse beschreven in dit document worden afgenomen

Binnen dit domein is er voortdurend sprake van technische vooruitgang. Daarom zouden wij, indien u hiermee akkoord gaat, het bacterieel genetisch materiaal geïsoleerd uit uw biologische stalen graag gedurende 25 jaar willen bewaren voor toekomstig onderzoek. Toekomstig onderzoek kan onder andere bestaan uit bijkomend onderzoek naar het genetische materiaal van de micro-organismen, met mogelijks nieuwere technieken, of onderzoek naar specifieke eigenschappen zoals stoffen geproduceerd door deze micro-organismen. Elk onderzoek buiten

de context die in dit document wordt beschreven, kan alleen plaatsvinden na goedkeuring van een ethisch comité.

Al het menselijk lichaamsmateriaal afkomstig van het Universitair Ziekenhuis Antwerpen (UZA) en de Universiteit Antwerpen zal verwerkt, gecodeerd en voor wetenschappelijke onderzoeksdoeleinden bewaard worden in de Biobank Antwerpen volgens het koninklijk besluit van 9 januari 2018.

## 7. Vertrouwelijkheid

Alle persoonsgegevens en informatie die u tijdens de studie zal aanleveren via de vragenlijsten zal vertrouwelijk worden behandeld. Daarnaast zal de verwerking van de door u aangeleverde persoonsgegevens verlopen conform de Algemene Verordening Gegevensbescherming (ook bekend als GDPR) en de relevante Belgische wetgeving¹. Tijdens het verloop van de studie zullen uw stalen en de bijhorende resultaten aan een persoonlijke code worden gekoppeld. Door te werken met pseudonimisering, waarbij uw persoonsgegevens via een code worden omgezet naar versleutelde gegevens, kunnen wij u in een latere fase persoonlijke feedback bezorgen over uw microbioomprofiel met extra duiding. De sleutel van de code tot de koppeling naar je persoonsgegevens is beveiligd met een wachtwoord en enkel ter beschikking van de verantwoordelijke arts, hoofdonderzoeker en uitvoerende onderzoekers. Voor het zorgvuldig bewaren van de stalen, werken we samen met het Universitair Ziekenhuis Antwerpen en de Biobank Antwerpen. Indien de resultaten van deze studie gepubliceerd worden in een rapport of wetenschappelijk tijdschrift of op eender welke andere manier openbaar worden gemaakt, zal u nooit bij naam worden genoemd.

In het kader van het faciliteren van wetenschappelijk onderzoek zullen wij de over u verzamelde informatie en persoonsgegevens verder verwerken. Wij garanderen hierbij dat deze aanvullende verwerkingen compatibel zijn met de oorspronkelijke doeleinden waarvoor de door u aangeleverde gegevens in het kader van deze studie werden verzameld. De verdere verwerking van de stalen en verzamelde informatie voor secundair wetenschappelijke onderzoek is mogelijk. Verder kan dit ook mogelijk vervolgonderzoek met meer (commerciële) praktische toepassingen omvatten zoals de ontwikkeling van nieuwe testmethoden en behandelingen. Hierbij zullen de gegevens steeds gepseudonimiseerd ingezet worden.

De UAntwerpen heeft een functionaris voor gegevensbescherming. Indien u vragen of bezorgheden heeft aangaande de bescherming van uw persoonlijke gegevens, kan u een schriftelijke vraag richten tot Koen Pepermans, Sint-Jacobstraat 2, 2000 Antwerpen, België of privacy@uantwerpen.be.

## Recht op informatie, inzage, correctie en schrapping

U heeft het recht om informatie te vragen over de procedures en het beschreven onderzoeksproject. Alle redelijke vragen voor informatie zullen beantwoord worden door de hoofdonderzoekers naar best vermogen. Als er belangrijke veranderingen zijn in de procedures, de risico's of de voordelen van deze studie dan wordt u op de hoogte gebracht. Verder heeft u

<sup>&</sup>lt;sup>1</sup>https://www.gegevensbeschermingsautoriteit.be/sites/privacycommission/files/documents/Wet Loi 30 07 2018.pdf

ook recht op inzage tot uw persoonlijke resultaten (vragenlijstgegevens en analyseresultaten). U heeft ook het recht om uw persoonlijke gegevens te corrigeren of schrappen. Dit kan u doen door schriftelijk (via e-mail of brief) contact op te nemen met de hoofdonderzoekers.

#### Contact

Als u bijkomende informatie wenst, maar ook in geval van problemen of als u zich zorgen maakt, kan u altijd contact opnemen met het studieteam via mail (<u>isala@uantwerpen.be</u>). Indien nodig, verwijzen wij u door naar de verantwoordelijke arts Prof. Dr. Veronique Verhoeven.

Als u vragen heeft met betrekking tot uw rechten als deelnemer aan de studie, kan u contact opnemen met de ombudsdienst in het UZA op het telefoonnummer: 03/821 31 60. Indien nodig kan de ombudsdienst u in contact brengen met het Ethisch Comité.

## Het Rufaida project:

## Impact van Ramadan vasten op het darm en vaginale microbioom

#### II. Geïnformeerde toestemming

#### Deelnemer

Ik verklaar dat ik geïnformeerd ben over de aard, het doel, de duur, de eventuele voordelen en risico's van de studie en dat ik weet wat van mij wordt verwacht. Ik heb kennisgenomen van het informatiedocument en de bijlagen ervan.

Ik heb voldoende tijd gehad om na te denken en met een door mij gekozen persoon, zoals mijn huisarts of een familielid, te praten.

Ik heb alle vragen kunnen stellen die bij me opkwamen en ik heb een duidelijk antwoord gekregen op mijn vragen.

Ik begrijp dat mijn deelname aan deze studie vrijwillig is en dat ik vrij ben mijn deelname aan deze studie stop te zetten zonder dat dit mijn relatie schaadt met het therapeutisch team dat instaat voor mijn gezondheid.

Ik begrijp dat er tijdens mijn deelname aan deze studie gegevens over mij zullen worden verzameld en dat de arts-onderzoeker en de opdrachtgever de vertrouwelijkheid van deze gegevens verzekeren overeenkomstig de Belgische wetgeving ter zake.

Ik stem in met de verwerking van mijn persoonlijke gegevens volgens de modaliteiten die zijn beschreven in de rubriek over het verzekeren van de vertrouwelijkheid (zie bijlage). Ik geef ook toestemming voor de overdracht naar en verwerking van mijn gecodeerde gegevens in andere landen dan België.

Ik ga ermee akkoord / Ik ga er niet mee akkoord (**doorhalen wat niet van toepassing is**) dat de studiegegevens die voor de hier vermelde studie worden verzameld, later zullen worden verwerkt, op voorwaarde dat deze verwerking beperkt blijft tot de context van de hier vermelde studie.

Ik ga ermee akkoord / Ik ga er niet mee akkoord (**doorhalen wat niet van toepassing is**) dat ik tijdens de studie op 8 tijdspunten vaginale en darmstalen afneem.

Ik ga ermee akkoord / Ik ga er niet mee akkoord (doorhalen wat niet van toepassing is) dat de opdrachtgever de tijdens de studie verzamelde biologische stalen gedurende 25 jaar bewaart voor latere analyses, op voorwaarde dat dit beperkt blijft tot de context van de hier vermelde studie

Ik ga ermee akkoord / Ik ga er niet mee akkoord (doorhalen wat niet van toepassing is) dat ik op het einde van de studie mijn persoonlijk microbioom profiel kan bekijken via een unieke webpagina op de Isala website.

Ik heb een exemplaar ontvangen van de informatie aan de deelnemer en de geïnformeerde toestemming.

| Naam en voornaam van de deelnemer: | |
|---|---|
| Geboortedatum:/ | |
| Ik heb het informatie- en toestemmingsformulier gelezen. Ik begrijp de voor van deze studie, maar ook de eventuele risico's. Ik begrijp dat ik binnen uitgebreide vragenlijst krijg om te bepalen welke factoren een effect zouder het microbioom. Ik neem vrijwillig deel aan deze studie. | het onderzoek een |
| / | |
| Handtekening (naam, voornaam) | Datum |

## Verklaring van de hoofdonderzoeker

De hoofdonderzoekers Prof. Dr. Veronique Verhoeven en Prof. Dr. Ir. Sarah Lebeer zijn verantwoordelijk om dit onderzoeksprogramma uit te voeren volgens de voorwaarden die beschreven zijn in dit document.

## Verantwoordelijke arts

Prof. Dr. Veronique Verhoeven, Departement Family Medicine and Population Health (FAMPOP), Doornstraat 331, 2610 Wilrijk (Antwerpen) Tel: 03/265 25 18

## Verantwoordelijke microbiologe

Prof. Dr. Ir. Sarah Lebeer, Faculteit Wetenschappen, Departement Bioingenieurswetenschappen, Campus Groenenborger, Groenenborgerlaan 171, 2020 Antwerpen Tel: 03/265 32 85

#### **Hoofdonderzoeker**

Ik ondergetekende Prof. Dr. Veronique Verhoeven, hoofdonderzoeker, verklaar de benodigde informatie inzake deze studie aan de deelnemer te hebben verstrekt evenals een exemplaar van het informatiedocument.

Ik bevestig dat geen enkele druk op de deelnemer is uitgeoefend om hem/haar te doen toestemmen tot deelname aan de studie en ik ben bereid om op alle eventuele bijkomende vragen te antwoorden.

Ik bevestig dat ik werk in overeenstemming met de ethische beginselen zoals vermeld in de laatste versie van de "Verklaring van Helsinki", de "Goede klinische praktijk" en de Belgische wet van 7 mei 2004 inzake experimenten op de menselijke persoon.

Handtekening hoofdonderzoeker: Datum: ...../.....

#### Hoofdonderzoeker

Ik ondergetekende Prof. Dr. Ir. Sarah Lebeer, hoofdonderzoeker, verklaar de benodigde informatie inzake deze studie aan de deelnemer te hebben verstrekt evenals een exemplaar van het informatiedocument.

Ik bevestig dat geen enkele druk op de deelnemer is uitgeoefend om hem/haar te doen toestemmen tot deelname aan de studie en ik ben bereid om op alle eventuele bijkomende vragen te antwoorden.

Ik bevestig dat ik werk in overeenstemming met de ethische beginselen zoals vermeld in de laatste versie van de "Verklaring van Helsinki", de "Goede klinische praktijk" en de Belgische wet van 7 mei 2004 inzake experimenten op de menselijke persoon.

Handtekening hoofdonderzoeker: Datum: ...../......

## Het Rufaida project:

Impact van Ramadan vasten op het darm en vaginale microbioom

## III. Aanvullende informatie over de bescherming en de rechten van deelnemers aan een klinische studie

#### Ethische comités

Deze studie werd geëvalueerd door een onafhankelijk ethisch comité UZA/UA dat een gunstig advies heeft uitgebracht. De ethische comités hebben als taak de personen die aan klinische studies deelnemen te beschermen. Ze controleren of uw rechten als patiënt en als deelnemer aan een studie gerespecteerd worden, of - uitgaande van de huidige kennis - de balans tussen risico's en voordelen gunstig is voor de deelnemers, of de studie wetenschappelijk relevant en ethisch verantwoord is.

Hierover brengen de ethische comités een advies uit in overeenstemming met de Belgische wet van 7 mei 2004. U dient het positief advies van de Ethische Comités in geen geval te beschouwen als een aansporing om deel te nemen aan deze studie.

#### Vrijwillige deelname

Aarzel niet om alle vragen te stellen die bij u opkomen voordat u tekent. Neem de tijd om er over te praten met een vertrouwenspersoon indien u dat wenst.

U heeft het recht om niet deel te nemen aan deze studie of met deze studie te stoppen, zonder dat u hiervoor een reden hoeft te geven, zelfs al hebt u eerder toegestemd om aan deze studie deel te nemen. Uw beslissing zal in geen geval uw relatie met de arts-onderzoeker beïnvloeden, noch de kwaliteit van uw verdere verzorging.

Als u aanvaardt om aan deze studie deel te nemen, ondertekent u het toestemmingsformulier. De arts-onderzoeker zal dit formulier ook ondertekenen en zal zo bevestigen dat hij u de noodzakelijke informatie over deze studie heeft gegeven. U zal het voor u bestemde exemplaar ontvangen.

Voor uw veiligheid is het wel aanbevolen om de arts-onderzoeker op de hoogte te stellen indien u besluit uw deelname aan de studie stop te zetten.

## Kosten in verband met uw deelname

Indien u besluit om aan deze studie deel te nemen, brengt dit dus geen bijkomende kosten met zich mee voor u of voor uw verzekeringsmaatschappij. De bezoeken en procedures die behoren tot deze studie en die vermeld worden in de beschrijving van het verloop van de studie op pagina 3 tot 4 of in de figuur op pagina 3 worden door de opdrachtgever betaald.

## Vertrouwelijkheidsgarantie

Uw deelname aan de studie betekent dat u ermee akkoord gaat dat de arts-onderzoeker gegevens over u verzamelt en dat de opdrachtgever van de studie die gebruikt voor onderzoek en in het kader van wetenschappelijke en medische publicaties.

U hebt het recht om aan de arts-onderzoeker te vragen welke gegevens hij/zij over u heeft verzameld en waarvoor ze gebruikt worden in het kader van de studie. Deze gegevens hebben betrekking op uw huidige klinische situatie maar ook op uw medische voorgeschiedenis en op de resultaten van onderzoeken die werden uitgevoerd voor de behandeling van uw gezondheid

volgens de geldende zorgstandaard. U hebt het recht om deze gegevens in te kijken en om verbeteringen te laten aanbrengen indien ze foutief zouden zijn<sup>2</sup>.

De arts-onderzoeker is verplicht om deze verzamelde gegevens vertrouwelijk te behandelen.

Dit betekent dat hij/zij zich ertoe verbindt om uw naam nooit bekend te maken bv. in het kader van een publicatie of een conferentie en dat hij/zij uw gegevens zal coderen (uw identiteit zal worden vervangen door een identificatiecode in de studie) voordat hij/zij ze doorgeeft aan de beheerder van de databank.

De arts-onderzoeker en zijn/haar team zullen gedurende de volledige studie de enige personen zijn die een verband kunnen leggen tussen de overgedragen gegevens en uw medisch dossier<sup>3</sup>.

De overgedragen persoonlijke gegevens omvatten geen combinatie van elementen waarmee het mogelijk is u te identificeren<sup>4</sup>.

De door de opdrachtgever aangestelde beheerder van de onderzoeksgegevens kan u niet identificeren op basis van de overgedragen gegevens. Deze persoon is verantwoordelijk voor het verzamelen van de gegevens die door alle artsen-onderzoekers die deelnemen aan de studie zijn verzameld en voor de verwerking en de bescherming van die gegevens in overeenstemming met de Belgische wet betreffende de bescherming van de persoonlijke levenssfeer.

Om de kwaliteit van de studie te controleren, kan uw medisch dossier worden ingekeken door personen die gebonden zijn aan het beroepsgeheim zoals vertegenwoordigers van de ethische comités, van de opdrachtgever van de studie of een extern auditbureau. Dit kan enkel gebeuren onder strikte voorwaarden, onder de verantwoordelijkheid van de arts-onderzoeker en onder zijn/haar toezicht (of van één van zijn/haar onderzoeksmedewerkers).

De (gecodeerde) onderzoeksgegevens kunnen doorgegeven worden aan Belgische of andere regelgevende instanties, aan de betrokken ethische comités, aan andere artsen en/of instellingen die samenwerken met de opdrachtgever.

Ze kunnen ook doorgegeven worden aan andere sites van de opdrachtgever in België en in andere landen waar de normen inzake de bescherming van persoonsgegevens verschillend of minder strikt kunnen zijn<sup>5</sup>. Dit gebeurt dan steeds in gecodeerde vorm zoals hierboven uitgelegd.

Uw toestemming om aan deze studie deel te nemen betekent dus ook dat u akkoord gaat dat uw gecodeerde medische gegevens gebruikt worden voor doeleinden die in dit informatieformulier beschreven staan en dat ze overgedragen worden aan bovenvermelde personen en/of instellingen.

De opdrachtgever zal de verzamelde gegevens gebruiken in het kader van de studie waaraan u deelneemt, maar wil ze ook kunnen aanwenden in het kader van andere studies. Buiten de

Informatie- en toestemmingsformulier – Versie 2 – 24 januari 2025

Pagina 12 van 14

<sup>&</sup>lt;sup>2</sup> Deze rechten zijn bepaald door de wet van 8 december 1992 tot bescherming van de persoonlijke levenssfeer ten opzichte van de verwerking van persoonsgegevens en door de wet van 22 augustus 2002 betreffende de rechten van de patiënt.

<sup>&</sup>lt;sup>3</sup> Voor klinische studies verplicht de wet om het verband met uw dossier gedurende 20 jaar te behouden. In geval van een studiegeneesmiddel voor een innoverende therapie waarbij gebruik wordt gemaakt van menselijk lichaamsmateriaal, bedraagt deze periode minimaal 30 jaar en maximaal 50 jaar in overeenstemming met de Belgische wet van 19 december 2008 inzaek het gebruik van menselijk lichaamsmateriaal en de geldende Koninklijke Besluiten.

<sup>&</sup>lt;sup>4</sup> De gegevensbank met onderzoeksresultaten bevat dus geen verband met elementen zoals uw initialen, uw geslacht en uw volledige geboortedatum (dd/mm.iiii).

<sup>&</sup>lt;sup>5</sup> De opdrachtgever verbindt zich er toe om de voorwaarden in de Europese Richtlijnen en de Belgische Wetgeving betreffende de bescherming van de persoonlijke levenssfeer te eerbiedigen.

context die beschreven wordt in dit document, kunnen uw gegevens enkel gebruikt worden als een ethisch comité haar goedkeuring heeft gegeven.

Indien u uw toestemming tot deelname aan de studie intrekt, zullen de gecodeerde gegevens die al verzameld waren vóór uw terugtrekking, bewaard worden. Hierdoor wordt de geldigheid van de studie gegarandeerd. Er zal geen enkel nieuw gegeven aan de opdrachtgever worden doorgegeven.

#### Wat gebeurt er met uw staal/stalen tijdens en na afloop van de studie<sup>6</sup>?

Voor de stalen wordt ook een coderingprocedure gebruikt net zoals voor uw medische gegevens. De aan de opdrachtgever overgedragen stalen zijn dus enkel voorzien van een identificatiecode in het kader van deze klinische studie.

De beheerder van deze stalen (Departement Bio-Ingenieurswetenschappen, Laboratorium voor Toegepaste Microbiologie en Biotechnologie, UAntwerpen) verbindt zich ertoe deze stalen alleen in het kader van deze klinische studie te gebruiken en ze te vernietigen na afloop van de voorziene bewaarperiode.

Het biologisch materiaal wordt beschouwd als een "gift" en u dient zich ervan bewust te zijn dat u in principe geen enkel financieel voordeel (royalties) zal ontvangen in verband met de ontwikkeling van nieuwe therapieën die voortvloeien uit het gebruik van het door u geschonken biologisch materiaal dat een commerciële waarde zou kunnen hebben.

Indien u uw toestemming tot deelname aan de studie intrekt, kan u uw staal/stalen laten vernietigen of terug opvragen. Neem daarvoor contact op met de arts-onderzoeker. De resultaten die op basis van uw staal/stalen werden verkregen voordat u uw toestemming tot deelname hebt ingetrokken, blijven eigendom van de opdrachtgever.

### Verzekering

Elke deelname aan een studie houdt een risico in, hoe klein ook. De opdrachtgever is - ook indien er geen sprake is van fout - aansprakelijk voor de schade die de deelnemer of in geval van overlijden zijn/haar rechthebbenden, oplopen en die rechtstreeks of onrechtstreeks verband houdt met diens deelname aan de studie. U moet hiervoor dus geen fout aantonen. De opdrachtgever heeft voor deze aansprakelijkheid een verzekering afgesloten<sup>7</sup>.

We verzoeken u daarom om elk nieuw gezondheidsprobleem aan de arts-onderzoeker te melden. Hij/Zij kan u aanvullende informatie verstrekken over mogelijke behandelingen.

Indien de arts-onderzoeker van mening is dat er een verband met de studie mogelijk is (er is geen verband met de studie bij schade ten gevolge van het natuurlijke verloop van uw ziekte of ten gevolge van gekende bijwerkingen van uw standaardbehandeling), zal hij/zij de opdrachtgever van de studie op de hoogte stellen die de aangifteprocedure bij de verzekering zal starten. Deze zal, indien zij het nodig acht, een expert aanstellen om een oordeel uit te spreken over het verband tussen uw nieuwe gezondheidsklachten en de studie.

In het geval van onenigheid met de arts-onderzoeker of met de door de verzekeringsmaatschappij aangestelde expert, en steeds wanneer u dit nodig acht, kunnen u of in geval van overlijden uw rechthebbenden de verzekeraar rechtstreeks in België dagvaarden.

<sup>&</sup>lt;sup>6</sup> In overeenstemming met artikel 29 van de Belgische Wet inzake experimenten op de menselijke persoon (7 mei 2004).

| De wet voorziet dat de dagvaarding van de verzekeraar kan gebeuren ofwel voor de rechter van de plaats waar de schadeverwekkende feiten zich hebben voorgedaan, ofwel voor de rechter van uw woonplaats, ofwel voor de rechter van de zetel van de verzekeraar. |
|---|
| van uw woonplaats, ofwer voor de reenter van de zeter van de verzekerdar. |
| Informatie- en toestemmingsformulier – Versie 2 – 24 januari 2025 Pagina 14 van 14 |